CLINICAL TRIAL: NCT05881889
Title: Effects of Repetitive Transcranial Magnetic Stimulation on Fear of Cancer Recurrence: mPFC-amygdala-hippocampus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8220053738
Record Dates: First submitted 2023-03-20; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-02

CONDITIONS: Psychology

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- repetitive transcranial magnetic stimulation (Experimental): For patients in the rTMS group, we will first determine the intensity of the rTMS protocol by assessing the individual resting motor threshold (rMT). After determination of each individual's rMT, we will set rTMS intensity at 100% of the rMT and apply a single train of low-frequency rTMS over the DLPFS at 1 Hz for a total duration of 30 min (2000 pulses). receive 4 week rTMS treatment.
  Interventions: Device: low-frequency repetitive transcranial magnetic stimulation
- sham stimulation (Sham Comparator): For patients in the sham group, we will apply rTMS over the DLPFS in sham modality.
  Interventions: Device: sham low-frequency repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: low-frequency repetitive transcranial magnetic stimulation — For patients in the rTMS group, we will first determine the intensity of the rTMS protocol by assessing the individual resting motor threshold (rMT). After determination of each individual's rMT, we will set rTMS intensity at 100% of the rMT and apply a single train of low-frequency rTMS over the DLPFS at 1 Hz for a total duration of 30 min (2000 pulses).
  Arms: repetitive transcranial magnetic stimulation
Device: sham low-frequency repetitive transcranial magnetic stimulation — sham low-frequency repetitive transcranial magnetic stimulation
  Arms: sham stimulation

SUMMARY:
Introduction: Previous studies have shown that many breast cancer patients are suffering from fear of cancer recurrence (FCR). However, effective physical intervention for FCR has been scarce. In this study, low-frequency repetitive transcranial magnetic stimulation (rTMS) targeting the right dorsolateral prefrontal cortex (DLPFC) will be applied on patients with high FCR. We aim to assess the efficacy of low-frequency rTMS in the treatment of FCR in breast cancer patients.

Methods and analysis: This will be a two-arm, randomised controlled trial comparing rTMS, sham stimulation in breast cancer patients with high FCR. A total of 50 breast cancer patients with a high FCR score (>27) will be recruited. Patients will be randomly assigned to receive 4-week rTMS, sham stimulation. Assessments will be conducted at week 0 (baseline), week 4 (the end of intervention), week 5 (1 week post-treatment), week 8 (1 month post-treatment), and week 16 (3 months post-treatment). The primary outcome of the study will be to ascertain, whether the rTMS program is sufficient in relieving FCR in breast cancer patients (measured by the 7-item FCR scale). Additionally, GAD7, PHQ9, NRS, and ISI7 will be used to measure individual's anxiety, depression, pain, and insomnia symptoms.

DETAILED DESCRIPTION:
This study will be a parallel assignment randomised controlled trial (RCT). Patients will be randomly assigned to rTMS intervention group (rTMS+ TAU), sham stimulation group (sham+ TAU). Treatment will be performed 5 times a week for 4 weeks. Assessments will be conducted at week 0 (baseline), week 4 (the end of intervention), week 5 (1 week post-treatment), week 8 (1 month post-treatment), and week 16 (3 months post-treatment). The screening, assessments, allocation and intervention will all be carried out via a WeChat mini Program (a widely used social communication application, with more than 1.2 billion users in China) specially tailored for the trial. An information sheet will be provided online, and informed consent will be completed online before participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult;
2. Breast cancer patients undergoing treatment for the first time;
3. Able to understand and sign informed consent;
4. Being able to comply with the intervention.

Exclusion Criteria:

1. Minors;
2. Having a diagnosis for a significant untreated mental or medical illness (e.g., consciousness disturbances, mania, acute phase of schizophrenia, major depressive disorder, etc.);
3. Patients with recurrent cancer;
4. Hospice patients.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Fear of Cancer Recurrence Questionnaire (FCRQ7) | we use FCRQ7 to assess the change of FCR level from baseline to 4, 5, 8, 16 weeks follow up
  There are 7 items scored on 5 levels, the total score of each item is summed up. The score above 27 indicates that the patient has significant fear, which requires certain psychological intervention and treatment.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ9) | we use PHQ9 to assess the change of depression level from baseline to 4, 5, 8, 16 weeks follow up
  The PHQ9 strictly conforms to the 9 symptomatic criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM5), with each item scoring 0-3 points and the total value range 0-27 points. PHQ9 can be used for both screening and evaluating the severity of depression. The results of PHQ9 are graded as follows: 0-4: no depression; 5-9: mild depression; 10-14: moderate depression; 15-19: moderate to severe depression; and 20-27: severe depression
Generalized Anxiety Disorder (GAD7) | we use GAD7 to assess the change of anxiety level from baseline to 4, 5, 8, 16 weeks follow up
  The total score is categorized as follows: 0-4: no generalized anxiety; 5-9: mild generalized anxiety; 10-14: moderate generalized anxiety; and 15-21: severe generalized anxiety.
Numeric Rating Scale (NRS) | we use NRS to assess the change of pain level from baseline to 4, 5, 8, 16 weeks follow up
  Participant's somatic pain level will be assessed using the "0-10" numeric rating scale (NRS) (i.e., how would you rate your pain at its worst over the past 3 days?) , in which 0 means 'no pain' and 10 means 'the worst pain'. Participants will be asked to select a number between 0 and 10, to indicate their current pain level. A total score of 4 or more indicates that the patient is currently suffering from pain.
Insomnia Severity Index (ISI) | we use ISI to assess the change of insomnia severity from baseline to 4, 5, 8, 16 weeks follow up
  The change in insomnia symptoms will be measured by the insomnia severity index (ISI) , which assesses the severity, nature, and impact of insomnia. It is a 7-item self-report measure, ranging from 0 (no problem) to 4 (very severe problem). The resulting sum score of the ISI ranges from 0 to 28. Higher scores indicate more severe insomnia symptoms.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu W, Zhao N, Li W, Qiu L, Luo X, Lin Y, Wang W, Garg S, Sun H, Yang Y. Effects of repetitive transcranial magnetic stimulation on fear of cancer recurrence and its underlying neuromechanism. Contemp Clin Trials Commun. 2024 Apr 23;39:101299. doi: 10.1016/j.conctc.2024.101299. eCollection 2024 Jun. PMID 38720913